CLINICAL TRIAL: NCT02786537
Title: THE PRIORITIZE STUDY: A Pragmatic, Randomized Study of Oral Regimens for Hepatitis C: Transforming Decision-Making for Patients, Providers, and Stakeholders
Brief Title: Study of Oral Treatments for Hepatitis C
Acronym: PRIORITIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Merck Sharp & Dohme LLC (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1234; PCORI-1503-27891 (Other: PCORI); IRB201501162 (Other: New UF IRB-01)
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir; ledipasvir; ledipasvir, sofosbuvir drug combination; Cytochrome P-450 CYP2B1; ombitasvir; dasabuvir; Viekira Pak; elbasvir; grazoprevir; elbasvir-grazoprevir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- EBR/GZR (elbasvir/grazoprevir) with RBV (Active Comparator): Patients received 1 EBR/GZR (elbasvir/grazoprevir) (Zepatier) tablet (50/100mg) once daily for 12 to 16 weeks (provider discretion) with Ribavirin (RBV) 200 mg/tablet, 1-3/day, taken 1-2 times per day (dosage at discretion of provider).
  Interventions: Drug: EBR/GZR (elbasvir/grazoprevir); Drug: Ribavirin
- EBR/GZR (elbasvir/grazoprevir) (Active Comparator): Patients received 1 EBR/GZR (elbasvir/grazoprevir) tablet (50/100 mg) once daily for 12 to 16 weeks (provider discretion) (without Ribavirin)
  Interventions: Drug: EBR/GZR (elbasvir/grazoprevir)
- SOF/LDV (sofosbuvir/ledipasvir) with RBV (Active Comparator): Patients received 1 SOF/LDV (sofosbuvir/ledipasvir) (Harvoni) tablet (400/90 mg) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (at discretion of provider). RBV taken as 200 mg/tablet(capsule), 1-3 pills/day, 1-2 times/day.
  Interventions: Drug: SOF/LDV (sofosbuvir/ledipasvir); Drug: Ribavirin
- SOF/LDV (sofosbuvir/ledipasvir) (Active Comparator): Patients received 1 SOF/LDV (sofosbuvir/ledipasvir) tablet (400/90 mg) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  Interventions: Drug: SOF/LDV (sofosbuvir/ledipasvir)
- PrOD (Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir) with RBV (Phase 1 only) (Active Comparator): Patients received Pr0D (Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir) orally daily with food for 12 to 24 weeks with RBV (Ribavirin). Ombitasvir/Paritaprevir/Ritonavir (12.5/75/50 mg/tablet) -2 tablets once daily with food for 12 to 24 weeks and 1 dasabuvir tablet (250 mg) twice daily with food for 12 to 24 weeks.
  RBV (200 mg/pill) 1-3 pills/day, 1-2 times/day (use and dosage at provider discretion). Total daily RBV dosage ranged from 200 to 1200 mg.
  Interventions: Drug: PrOD (ombitasvir/paritaprevir/ritonavir with dasabuvir) (Phase 1 only)
- PrOD (ombitasvir/paritaprevir/ritonavir and dasabuvir) (Active Comparator): Patients received 2 ombitasvir/paritaprevir/ritonavir tablets (12.5/75/50 mg) once daily and 1 dasabuvir (250 mg) tablet twice daily with food for 12 to 24 weeks without Ribavirin (as per provider instructions)
  Interventions: Drug: PrOD (ombitasvir/paritaprevir/ritonavir with dasabuvir) (Phase 1 only); Drug: Ribavirin

INTERVENTIONS:
Drug: SOF/LDV (sofosbuvir/ledipasvir) — Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
  Other Names: Harvoni® (sofosbuvir/ledipasvir)
  Arms: SOF/LDV (sofosbuvir/ledipasvir); SOF/LDV (sofosbuvir/ledipasvir) with RBV
Drug: PrOD (ombitasvir/paritaprevir/ritonavir with dasabuvir) (Phase 1 only) — Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) (2 tablets taken orally) and Dasabuvir (250 mg tablet) (1 tablet twice daily) with food for 12 to 24 weeks (treatment duration as per HCV provider)
  Other Names: Viekira Pak/Viekira
  Arms: PrOD (Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir) with RBV (Phase 1 only); PrOD (ombitasvir/paritaprevir/ritonavir and dasabuvir)
Drug: EBR/GZR (elbasvir/grazoprevir) — Elbasvir/grazoprevir (50/100mg) tablet once daily with or without food with or without RBV for 12 to 16 weeks
  Other Names: Zepatier
  Arms: EBR/GZR (elbasvir/grazoprevir); EBR/GZR (elbasvir/grazoprevir) with RBV
Drug: Ribavirin — 200 mg pills (1-3 pills, 1-2 times per day)
  Other Names: RBV
  Arms: EBR/GZR (elbasvir/grazoprevir) with RBV; PrOD (ombitasvir/paritaprevir/ritonavir and dasabuvir); SOF/LDV (sofosbuvir/ledipasvir) with RBV

SUMMARY:
Phase 1 of this study compared the effectiveness of 3 approved DAA (direct-acting antiviral) HCV treatment regimens to learn whether they worked equally well under real-world conditions. Phase 2 of this study began early 2017 with removal of 1 DAA regimen, limiting randomization to just 2 FDA approved DAA regimens. Patients receiving HCV therapy in community and academic clinics were offered the opportunity to consent to be randomly assigned to one of three (phase 1) or one of two (phase 2) regimens and observed for outcomes. Once randomized, all medical care, laboratory testing, and any disease or side effect management were assumed by usual care conditions, and patient-reported outcomes were collected outside clinic in keeping with pragmatic design principles.

DETAILED DESCRIPTION:
In Phase 1 of this study, consented patients were randomized to 1 of the following 3 HCV DAA treatments: 1) Harvoni® (SOF/LDV) 2) Viekira Pak™ (PrOD) 3) Zepatier™ (EBR/GZR) with the optional addition of Ribavirin (RBV) and the length of treatment determined by the individual provider.

In Phase 2 of this study, consented patients were randomized to 1 of 2 FDA approved HCV treatments: Harvoni® or Zepatier™. Both Phase 1 and Phase 2 subjects had up to 1 tablespoon of blood drawn for HCV resistance testing and future biorepository testing (following appropriate additional consent). The results of testing determined whether a genotype 1a subject randomized to Zepatier would be provided 12 or 16 wks of Zepatier.

Following enrollment/randomization, participants completed patient reported outcome questionnaires (PROs) via electronic device or telephone. Following baseline/randomization, participants were asked to complete surveys again at Wk 4 of treatment, End of Treatment, 1 and 3 year post treatment. Patients continued standard medical care throughout study. Data was abstracted from test results and medical records throughout treatment and for up to 3 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCV Genotype 1a or 1b
* Adult patients (age 18 years or older)
* Patients being prescribed HCV treatment who can begin treatment with any of the three HCV treatments being studied (Harvoni (SOF/LDV), Viekira Pak (PrOD) (Phase 1 only), or Zepatier (EBR/GZR))

Exclusion Criteria:

* Inability to provide written informed consent
* HARVONI® is not a covered drug on benefits formulary
* Current or historical evidence of hepatic decompensation (variceal bleeding, hepatic encephalopathy, or ascites)
* Child Pugh (CTP) B or C Cirrhosis (documented CTP calculation is required)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06-13 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Nelson, MD, Principal Investigator — University of Florida
Locations (37):
- United States (37):
  - Liver Wellness Center, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - UCSD Medical Center, San Diego, California
  - UCSF/Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - Univ of California, San Francisco, San Francisco, California
  - Yale University Digestive Diseases, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - University of Miami/Schiff Center for Liver Diseases, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Internal Medicine Associates of Wellstar Atlanta Medical Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - John Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - GI Associates & Endoscopy Center, Flowood, Mississippi
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Ctr, Omaha, Nebraska
  - Southwest CARE Center, Santa Fe, New Mexico
  - Mt. Sinai Beth Israel, New York, New York
  - New York Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mountain View Medical Center, Valatie, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Research Specialist of Texas, Houston, Texas
  - Bon Secours St. Mary 's Hospital of Richmond (Liver Institute of Virginia), Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evon DM, Dong M, Reeve BB, Peter J, Michael L, Lok AS, Nelson DR, Stewart PW. Sustainable and equivalent improvements in symptoms and functional well-being following viral cure from ledipasvir/sofosbuvir versus elbasvir/grazoprevir for chronic hepatitis C infection: Findings from the randomized PRIORITIZE trial. J Viral Hepat. 2022 Sep;29(9):795-806. doi: 10.1111/jvh.13716. Epub 2022 Jun 15. PMID 35657133
- [Derived] Lok AS, Moon J, Sherman KE, Khalili M, Fishbein D, Reddy KR; PRIORITIZE Study Team. Long-term Follow-up of Hepatitis C Patients Who Achieved Sustained Virologic Response in the Pragmatic PRIORITIZE Study. Clin Gastroenterol Hepatol. 2023 Feb;21(2):546-548.e4. doi: 10.1016/j.cgh.2022.01.059. Epub 2022 Feb 17. PMID 35182741
- [Derived] Sulkowski MS, Moon JS, Sherman KE, Morelli G, Darling JM, Muir AJ, Khalili M, Fishbein DA, Hinestrosa F, Shiffman ML, Di Bisceglie A, Rajender Reddy K, Pearlman B, Lok AS, Fried MW, Stewart PW, Peter J, Wadsworth S, Kixmiller S, Sloan A, Vainorius M, Horne PM, Michael L, Dong M, Evon DM, Segal JB, Nelson DR; PRIORITIZE Study Team. A Pragmatic, Randomized Controlled Trial of Oral Antivirals for the Treatment of Chronic Hepatitis C: The PRIORITIZE Study. Hepatology. 2021 Dec;74(6):2952-2964. doi: 10.1002/hep.32053. Epub 2021 Aug 26. PMID 34255381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consented at 34 US centers Between June 2016 and March 2018. Patients' insurance was screened for inclusion of SOF/LDV on formulary (the HCV regimen not provided by the study). However, following randomization, participants who were unable to obtain SOF/LDV through insurance received 1 of 2 Direct Acting Antiviral (DAA) HCV Treatment regimens 1)EBR/GZR or 2)PrOD during Phase 1 and received EBR/GZR during Phase 2.
Pre-assignment Details: This study initially (Phase 1) randomized subjects to receive 1 of 3 HCV DAA regimens (EBR/GZR +/- RBV, LDV/SOF +/- RBV, or PrOD +/-RBV). In phase 2 of this study, randomization to PrOD regimen was discontinued and newly enrolled subjects were randomized to either EBR/GZR +/- RBV or LDV/SOF +/- RBV. Efficacy data was analyzed via original 'randomization' and as subjects were 'actually treated (regimen actually received)' while safety analysis was evaluated by actual treatment received.
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) (Zepatier™) orally once daily with RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food and with RBV: Ribavirin (200 mg pill) 1-3 pills/day, once or twice daily. Total daily dosage ranged from 200 to 1200 mg.
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) (Zepatier™) orally once daily (without RBV) for 12 to 16 weeks
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks. Duration of treatment according to HCV treatment provider.
- SOF/LDV With RBV: Patients received SOF/LDV(sofosbuvir/ledipasvir) (Harvoni®) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV/sofosbuvir/ledipasvir: Sofosbuvir/Ledipasvir (400/90 mg) 1 tablet daily for approximately 12 to 24 weeks (treatment duration is per discretion of HCV provider) RBV (200 mg pill): 1-3 pills, once or twice daily (dosing per discretion of HCV provider). Total daily dosage ranged from 200 to 1200 mg.
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) (Harvoni®) orally once daily with or without food 12 to 24 weeks
  SOF/LDV: Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks (treatment duration is per discretion of HCV provider)
- PrOD/RBV(Phase 1 Only): PrOD: Two ombitasvir/paritaprevir/ritonavir once daily and dasabuvir (Viekira) once or twice daily with a meal for 12 to 24 weeks + RBV (provider discretion). Randomization to PrOD discontinued January 2017.
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks with food (treatment duration and use of ribavirin as per HCV provider)
  Dasabuvir: 250 mg twice daily for 12 to 24 weeks with a meal RBV: Ribavirin 200 to 600 mg once or twice daily
- PrOD (Phase 1 Only): Randomization to Prod discontinued January 2017 (defining end of Phase 1) PrOD: Two ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily for 12 to 24 weeks
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks (treatment duration as per HCV provider)
  Dasabuvir: 250 mg daily for 12 to 24 weeks
Period: As Randomized
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD/RBV(Phase 1 Only) | PrOD (Phase 1 Only)
Started | 56 | 644 | 15 | 413 | 99 | 48
Completed | 50 | 582 | 15 | 378 | 87 | 41
Not Completed | 6 | 62 | 0 | 35 | 12 | 7
Not completed — Adverse Event | 0 | 11 | 0 | 4 | 6 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 2 | 0 | 3 | 1 | 0
Not completed — Non-compliance with study drug | 1 | 11 | 0 | 1 | 0 | 1
Not completed — Lost to treatment follow-up | 4 | 32 | 0 | 24 | 4 | 4
Not completed — Incarceration | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Opiate Dependency Relapse | 0 | 1 | 0 | 0 | 0 | 0
Not completed — HCV drugs stolen from pt | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Advised to stop after lapse in dosing | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject lost insurance | 0 | 0 | 0 | 1 | 0 | 0
Period: As Treated
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD/RBV(Phase 1 Only) | PrOD (Phase 1 Only)
Started (Numbers represent treatment regimen that study participant actually started (received).) | 56 | 664 | 15 | 394 | 99 | 47
Completed | 50 | 602 | 15 | 359 | 87 | 40
Not Completed | 6 | 62 | 0 | 35 | 12 | 7
Not completed — Adverse Event | 0 | 11 | 0 | 4 | 6 | 2
Not completed — Death | 0 | 2 | 0 | 3 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 32 | 0 | 25 | 4 | 4
Not completed — Non-compliance with study drug | 1 | 11 | 0 | 1 | 0 | 1
Not completed — Lost insurance | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Incarceration | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Opiate dependency relapse | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Drugs stolen from patient | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Advised to stop tx after loss of meds | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study participants as randomized to HCV treatment
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) tablet tablet once daily with RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir 50/100mg tablet) once daily with or without food with or without RBV for 12 to 16 weeks (with RBV)
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) tablet tablet once daily without RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir 50/100mg tablet): 1 tablet once daily with or without food with or without RBV for 12 to 16 weeks (without RBV)
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  sofosbuvir/ledipasvir: Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks with Ribavirin (RBV) (treatment duration and use of ribavirin is per discretion of HCV provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (per discretion of provider)
  SOF/LDV: Sofosbuvir/Ledipasvir (400/90 mg tablet ) 1 tablet orally once daily for approximately 12 to 24 weeks
- PROD With RBV (Phase 1 Only): Phase 1 only - Two ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily for 12 to 24 weeks +/- RBV (provider discretion)
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks (treatment duration and use of ribavirin as per HCV provider)
  Dasabuvir: 250 mg daily for 12 to 24 weeks
- PROD (Phase 1 Only): Phase 1 only - Two ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily for 12 to 24 weeks
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks Dasabuvir: 250 mg daily for 12 to 24 weeks
- Total: Total of all reporting groups
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PROD With RBV (Phase 1 Only) | PROD (Phase 1 Only) | Total
Number analyzed (Participants) | 56 | 644 | 15 | 413 | 99 | 48 | 1275
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 547 | 8 | 319 | 86 | 35 | 1039
  >=65 years | 12 | 97 | 7 | 94 | 13 | 13 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.0) | 53.3 (12.2) | 61.1 (6.6) | 56.2 (11.1) | 54.5 (11.3) | 59.9 (10.1) | 54.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 280 | 6 | 157 | 35 | 16 | 507
  Male | 43 | 364 | 9 | 256 | 64 | 32 | 768
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 44 | 0 | 26 | 5 | 1 | 81
  Not Hispanic or Latino | 51 | 586 | 14 | 375 | 90 | 45 | 1161
  Unknown or Not Reported | 0 | 14 | 1 | 12 | 4 | 2 | 33
Region of Enrollment [Number; unit: participants]
  United States | 56 | 644 | 15 | 413 | 99 | 48 | 1275
HCV RNA [Mean (Standard Deviation); unit: 10^6 units IU/mL] | 4.9 (6.7) | 3.1 (4.9) | 5.9 (4.7) | 3.5 (4.4) | 3.5 (3.8) | 3.7 (4.2) | 3.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR12) mITT With Imputation-Phase 1 and 2 EBR/GZR, SOF/LDV
Description: SVR (Sustained Virologic Response) 12 will be defined as undetectable hepatitis C virus (HCV) RNA at 12 week follow-up visit (12 -24 weeks after HCV treatment discontinuation at discretion of provider).
  mITT with imputation (missing=failure). Total number of subjects reflects participants from EBR/GZR with or without RBV and SOF/LDV with or without RBV randomized during Phase 1 and Phase 2.
Time Frame: 12 weeks post-treatment
Population: mITT with imputation, Missing SVR data = Failure. Numbers represent participants according to arm randomized (Period 1). Population excludes participants who did not start any HCV treatment.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- EBR/GZR: Patients received EBR/GZV tablet (elbasvir/grazoprevir) once daily for 12 to 16 weeks
  EBR/GZV (50/100mg) tablet: once daily with or without food 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily (with or without food) for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 56 | 644 | 15 | 413
Participants | 40 | 516 | 14 | 335

2. Primary Outcome: Phase 1/2 Number of Participants With Sustained Virologic Response (SVR12-mITT Without Imputation)
Description: SVR (Sustained Virologic Response) 12 will be defined as undetectable hepatitis C virus (HCV) RNA at 12 week follow-up visit (12 -24 weeks after HCV treatment discontinuation as dictated by standard of care at each individual site).
  Number of subjects reflects participants who started EBR/GZR or SOF/LDV- based treatment (with or without RBV) during Phase 1 and 2.
Time Frame: 12-24 weeks post HCV treatment
Population: All mITT without imputation (missing data excluded). Includes only number of participants for whom SVR12 data is available and based on study drug as randomized (Period 1). Participants for whom SVR 12 is not available are excluded from this table.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR With RBV: Patients received elbasvir/grazoprevir (EBR/GZR) tablet orally once daily with or without Ribavirin (RBV) for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks Ribavirin (RBV) (200 mg pill)- 1-3 pills orally once or twice daily (dosage at provider discretion)
- EBR/GZR: Patients received elbasvir/grazoprevir (EBR/GZR) once daily for 12 to 16 weeks EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (treatment duration per discretion of provider)
  sofosbuvir/ledipasvir: 1 Sofosbuvir/Ledipasvir (400/90 mg) tablet once daily with or without food for approximately 12 to 24 weeks Ribavirin (200 mg pill): 200 to 600 mg once or twice daily (treatment duration and dosage of ribavirin as per discretion of HCV provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily for 12 to 24 weeks (treatment duration as per discretion of HCV treatment provider) SOF/LDV (400/90 MG TABLET): 1 tablet orally once daily for 12 to 24 weeks
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 46 | 540 | 15 | 344
Participants | 40 | 516 | 14 | 335

3. Primary Outcome: Phase 1-Sustained Virologic Response (SVR12) mITT With Imputation
Description: SVR (Sustained Virologic Response) 12 will be defined as patients who have undetectable hepatitis C virus (HCV) RNA at 12 week follow-up visit (12 -24 weeks after HCV treatment discontinuation as dictated by standard of care at each individual site).
  mITT with imputation (missing=failure). Total number of subjects reflects participants from Phase 1 only.
Time Frame: 12 weeks post-treatment
Population: mITT with imputation, Missing SVR data =failure. Numbers represent participants according to arm randomized (period 1). Population excludes participants who did not start any HCV treatment.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR: Patients received EBR/GZR tablet (elbasvir/grazoprevir) once daily for 12 to 16 weeks
  EBR/GZR (50/100mg) tablet: 1 tablet once daily with or without food 12 to 16 weeks
- PrOD With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV)
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily with food for 12 to 24 weeks (treatment duration and use of ribavirin as per HCV provider)
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily with food for 12 to 24 weeks (dosage at discretion of provider)
  RBV (200 mg tablet): 1-3 tablets once or twice daily for 12 to 24 weeks (dosage and duration at discretion of provider)
- PrOD: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks (treatment duration as per HCV provider)
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 13 | 134 | 6 | 105 | 99 | 48
Participants | 9 | 108 | 6 | 88 | 77 | 42

4. Primary Outcome: Phase 1 Number of Participants With Sustained Virologic Response (SVR12-mITT Without Imputation)
Description: SVR (Sustained Virologic Response) 12 will be defined as undetectable hepatitis C virus (HCV) RNA at 12 week follow-up visit (12 -24 weeks after HCV treatment discontinuation as dictated by standard of care at each individual site).
  Number of subjects reflects participants randomized during Phase 1 only.
Time Frame: 12 -24 weeks post-treatment
Population: Participants analyzed based on HCV treatment as assigned by randomization.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) tablet tablet once daily with Ribavirin (RBV) for 12 to 16 weeks (provider discretion)
  EBR/GZR: Elbasvir/grazoprevir (50/100mg) 1 tablet once daily with or without food with or without RBV for 12 to 16 weeks
  Ribavirin at dosages ranging from 200mg to 600 mg daily (or twice daily) can be added to HCV DAA treatment regimen at discretion of HCV treatment provider
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) tablet tablet once daily without RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR: 1 Elbasvir/grazoprevir (50/100mg) tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) tablet orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  sofosbuvir/ledipasvir: Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
  RBV: At discretion of provider, 200 mg pill, 1-3 pills/day, 1-2 times/day (daily dosing ranging from 200mg to 1200 mg daily) added to HCV treatment regimen
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (Sofosbuvir/Ledipasvir 400/90 mg tablet): 1 tablet daily for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
- PrOD With RBV: Patients received PrOD (ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily) for 12 to 24 weeks with Ribavirin (RBV) (use and dosage at provider discretion)
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet ) 2 tablets daily for 12 to 24 weeks (treatment duration and use of ribavirin as per HCV provider) Dasabuvir: 500 mg tablet once or twice daily (morning and evening)
  RBV: At discretion of provider, 200 mg pill, 1-3 pills/day, 1-2 times/day (daily dosing ranging from 200mg to 1200 mg daily) added to HCV treatment regimen
- PrOD (Phase 1 Only): Patients received ProD (ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily) for 12 to 24 weeks without Ribavirin (at provider discretion)
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks (treatment duration and use of ribavirin as per HCV provider)
  Dasabuvir: 250 mg tablet twice daily for 12 to 24 weeks
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD (Phase 1 Only)
Number analyzed (Participants) | 10 | 113 | 6 | 92 | 80 | 42
Participants | 9 | 108 | 6 | 88 | 77 | 42

5. Primary Outcome: Mean Change in Headache-PRO Scores -Phase 1
Description: Headache was evaluated by the HIT-6 score, a validated, Patient Reported Outcomes survey (PROs) 'PROMIS Headache Impact Test (HIT)' with scores ranging from 36 to 78 with higher score reflecting greater impact. Mean change in headache side effect was evaluated using difference between baseline value of HIT-6 score to the highest (worst) score during treatment. Estimates of mean change and differences obtained from a constrained longitudinal linear mixed-effects model that treated baseline score as one of outcomes. Negative values for mean change represent improvement in symptom.
Time Frame: Baseline to On-Treatment
Population: Analysis limited to patients who completed a baseline and on-treatment PRO and as treated (Period 2) during Phase 1 only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With Ribavirin (RBV): Patients received EBR/GZR (elbasvir/grazoprevir) once daily withRBV (at discretion of provider) for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg - 1 tablet once daily with or without food for 12 to 16 weeks RBV: Ribavirin (200 mg pills) 1-3 pills/day, 1-2 times/day (Total dosage 200-1200 mg day)
- EBR/GZR Regimen: Patients received EBR/GZR (elbasvir/grazoprevir) once daily without RBV (at discretion of provider) for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg - 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with ribavirin (RBV)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) without ribavirin (RBV)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
- PrOD With RBV Regimen: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  RBV (200 mg pill): 1-3 pills once or twice daily for 12 to 24 weeks (dosage and duration at discretion of provider)
- PrOD: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks without Ribavirin (RBV). Treatment duration as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
Arm/Group | EBR/GZR With Ribavirin (RBV) | EBR/GZR Regimen | SOF/LDV With RBV | SOF/LDV | PrOD With RBV Regimen | PrOD
Number analyzed (Participants) | 9 | 84 | 5 | 61 | 62 | 28
units on a scale | 0.0 (1.4) | -0.8 (3.5) | -0.7 (5.0) | -0.5 (4.8) | -0.2 (4.7) | -2.2 (4.1)
Statistical Analysis 1: Comparison: SOF/LDV vs PrOD; PROD vs. SOF/LDV based regimens as reported in PRO (ALL PATIENTS WHO STARTED TREATMENT BY ARM AS TREATED), population limited to as randomization date of the last PrOD patient start date - RBV FREE REGIMENS; Test type: Superiority — Superiority test derived by comparing whether the 95% CI includes zero; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3.6 to 0.3] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method
Statistical Analysis 2: Comparison: EBR/GZR Regimen vs PrOD; RBV free EBR/GZR regimen compared to PrOD in consideration that RBV usage was determined by provider and not study randomization; Test type: Superiority; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.4 to 3.1] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method. CI for median derived from PROC QUANTREG

6. Primary Outcome: Mean Change in Headache-EBR/GZR and SOF/LDV
Description: Headache was evaluated by the HIT-6 score, a validated, Patient Reported Outcomes survey (PROs) 'PROMIS Headache Impact Test (HIT)' with scores ranging from 36 to 78 with higher score reflecting greater impact. Mean change in headache side effect was evaluated using difference between baseline value of HIT-6 score to the highest (worst) score during treatment. Estimates of mean change and differences obtained from a constrained longitudinal linear mixed-effects model that treated baseline score as one of outcomes. Negative values for mean change represent improvement, while negative values for 'difference' indicate LDV/SOF performed better than PrOD
Time Frame: Baseline to On-Treatment
Population: Analysis limited to participants who completed both baseline and end of treatment PRO
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg to 600mg tablet): 1 to 3 tablets once or twice daily (dosage and duration per discretion of provider)
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir ) once daily for 12 to 16 weeks (duration of treatment per provider discretion) without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 40 | 403 | 10 | 222
units on a scale | -0.8 (3.1) | -0.7 (4.4) | 0.4 (6.2) | -0.8 (5.0)
Statistical Analysis 1: Comparison: EBR/GZR vs SOF/LDV; Analysis based on RBV free EBR/GZR regimen vs SOF/LDV (all patients who started treatment by arm as treated); Test type: Superiority — Superiority test completed by comparing whether the 95% CI includes zero; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.6 to 1.0] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

7. Primary Outcome: Median Change in Headache -Phase 1
Description: Headache was evaluated by the HIT-6 score, a validated, Patient Reported Outcomes survey (PROs) 'PROMIS Headache Impact Test (HIT)' with scores ranging from 36 to 78 with higher score reflecting greater impact. Median change in headache side effect was evaluated using difference between baseline value of HIT-6 score to the highest (worst) score during treatment. Estimates of mean change and differences obtained from a constrained longitudinal linear mixed-effects model that treated baseline score as one of outcomes. Negative values for change represent improvement, while negative values for 'difference' indicate LDV/SOF performed better than PrOD
Time Frame: 12 weeks (Baseline and Average On-treatment Score)
Population: Analysis limited to patients randomized up to last patient randomized to PrOD and participants who completed baseline and on-treatment survey.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EBR/GZR (Elbasvir/Grazoprevir) With RBV: Patients received 1 EBR/GZR (elbasvir/grazoprevir) (Zepatier) tablet (50/100mg) once daily for 12 to 16 weeks (provider discretion) with Ribavirin (RBV)
  EBR/GZR (elbasvir/grazoprevir): Elbasvir/grazoprevir (50/100mg) tablet once daily with or without food with or without RBV for 12 to 16 weeks
  Ribavirin: 200 mg/tablet, 1-3/day, taken 1-2 times per day (dosage at discretion of provider).
- EBR/GZR (Elbasvir/Grazoprevir): Patients received 1 EBR/GZR (elbasvir/grazoprevir) tablet (50/100 mg) once daily for 12 to 16 weeks (treatment duration per provider discretion)
  EBR/GZR (elbasvir/grazoprevir): Elbasvir/grazoprevir (50/100mg) tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV (Sofosbuvir/Ledipasvir) With RBV: Patients received 1 SOF/LDV (sofosbuvir/ledipasvir) (Harvoni) tablet (400/90 mg) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (duration and usage of RBV at discretion of provider).
  SOF/LDV (sofosbuvir/ledipasvir): Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks
  Ribavirin (RBV): 200 mg/tablet(capsule), 1-3 pills/day, 1-2 times/day.
- SOF/LDV (Sofosbuvir/Ledipasvir): Patients received 1 SOF/LDV (sofosbuvir/ledipasvir) tablet (400/90 mg) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (sofosbuvir/ledipasvir): Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks (treatment duration at discretion of HCV provider)
Arm/Group | EBR/GZR (Elbasvir/Grazoprevir) With RBV | EBR/GZR (Elbasvir/Grazoprevir) | SOF/LDV (Sofosbuvir/Ledipasvir) With RBV | SOF/LDV (Sofosbuvir/Ledipasvir) | PrOD (Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir) With RBV (Phase 1 Only) | PrOD (Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir)
Number analyzed (Participants) | 9 | 84 | 5 | 61 | 62 | 28
units on a scale | 0.0 [-2.0 to 2.0] | 0.0 [-12.5 to 9.5] | -2.0 [-6.5 to 5.0] | -1.0 [-12.8 to 13.5] | 0.0 [-17.0 to 8.5] | -1.0 [-15.0 to 3.0]

8. Primary Outcome: Median Change in Headache-Phase 2
Description: Headache was evaluated by the HIT-6 score, a validated, Patient Reported Outcomes survey (PROs) 'PROMIS Headache Impact Test (HIT)' with scores ranging from 36 to 78 with higher score reflecting greater impact. Median change in headache side effect was evaluated using difference between baseline value of HIT-6 score to the highest (worst) score during treatment. Estimates of median change and differences obtained from a constrained longitudinal linear mixed-effects model that treated baseline score as one of outcomes. Negative values for mean change represent improvement, while negative values for 'difference' indicate LDV/SOF performed better than PrOD
Time Frame: Baseline -on Treatment (12-16 weeks)
Population: Analysis limited to patients randomized to EBR/GZR regimen or SOF/LDV regimen and participants who completed both baseline and on treatment survey.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV for 12 to 16 weeks.
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- EBR/GZR: Patients received EBR/GZR tablet (elbasvir/grazoprevir) once daily for 12 to 16 weeks (duration per investigator's discretion)
  EBR/GZR (50/100mg) tablet: 1 tablet once daily with or without food 12 to 16 weeks
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) without RBV
  SOF/LDV (400/90 mg tablet): 1 tablet once daily (with or without food) for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 40 | 403 | 10 | 222
units on a scale | -1.0 [-7.0 to 6.0] | 0.0 [-20.0 to 14.0] | 0.5 [-9.5 to 11.5] | -0.5 [-20.0 to 14.0]
Statistical Analysis 1: Comparison: EBR/GZR vs SOF/LDV; Analysis of EBR/GZR vs. SOF/LDV irrespective of RBV usage in consideration that RBV usage was determined by provider and not study randomization; Test type: Superiority — Superiority test comparison based on whether the 95% CI includes zero; Mean Difference (Net) = 0.5, 95% CI 2-sided [0.0 to 1.0] — The comparisons between regimens can be viewed as superiority test, by comparing whether the 95% CI includes zero

9. Primary Outcome: Mean Change in Nausea/Vomiting PRO Score -Phase 1
Description: Patients completed the PROMIS® Nausea Short Form at Baseline (T1) and on-treatment. PROMIS raw scores from each of the completed questionnaires were converted to standardized T-scores. Change was calculated as the difference between baseline and on-treatment score. T-scores for the PROMIS Nausea and Vomiting 4a scale range from 45.0 - 80.1. Higher scores indicate worse nausea. Negative values for mean change represent improvement.
  The estimates of mean change and differences were obtained from a constrained longitudinal linear mixed-effects model that treated the baseline score as one of the outcomes. The model expressed mean score as a function of DAA regimen, cirrhosis status, HCV genotype, sex, age, race, and previous treatment status.
Time Frame: Baseline to On-Treatment
Population: Analysis is limited to patients who completed at least one baseline and one end of treatment PRO survey during Phase 1 (end date corresponds to last PrOD patient start date)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir ) once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg to 600mg tablet): 1 to 3 tablets once or twice daily (dosage and duration per discretion of provider)
- PrOD With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- PrOD: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks without Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 8 | 79 | 5 | 58 | 59 | 25
units on a scale | 1.3 (5.0) | -1.4 (8.8) | -3.9 (4.0) | -0.7 (10.7) | 2.5 (8.6) | 0.7 (12.1)
Statistical Analysis 1: Comparison: SOF/LDV vs PrOD; Analysis based on RBV free SOF/LDV vs. PrOD in consideration that RBV usage was determined by provider and not study randomization and limited RBV sample size; Test type: Superiority — Superiority test comparison based on whether the 95% CI includes zero; Mean Difference (Net) = 1.4, 95% CI 2-sided [-4.2 to 7.0] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method
Statistical Analysis 2: Comparison: SOF/LDV vs PrOD; RBV free PrOD vs. SOF/LDV regimens (all patients who started treatment by arm as treated, population is limited to as randomization date of the last PrOD patient start date); Test type: Superiority — Superiority test comparison based on whether the 95% CI includes zero; Mean Difference (Net) = 1.4, 95% CI 2-sided [-4.2 to 7.0] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

10. Primary Outcome: Mean Change in Nausea/Vomiting PROMIS Score -EBR/GZR vs. LDV/SOF
Description: Participants completed the Patient Reported Outcomes surveys (PROs) 'PROMIS Nausea/Vomiting -4 Short Form' at baseline and during treatment. Raw scores are converted to standardized T-scores with a range of 45.0-80.1. Higher scores indicate worse nausea/vomiting.
  Results presented as mean difference from baseline to average of on Treatment Scores (highest/worst) score during treatment.
  A negative (-) PROMIS change score is suggestive of symptom improvement or lack of drug side effect. Estimates of mean change were obtained from a constrained longitudinal linear mixed-effects model that treated the baseline score as one of the outcomes.
Time Frame: Baseline and Average On-Treatment Score
Population: Patients with Baseline PROMIS Nausea/vomiting score who started treatment by arm as treated and completed baseline and on-treatment survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg tablet): 1 to 3 tablets once or twice daily (dosage and duration per discretion of provider)
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received 1 tablet SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage 200 mg- 1200 mg.
- SOF/LDV: Patients received 1 tablet SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 37 | 381 | 9 | 202
units on a scale | -0.3 (8.3) | -0.6 (8.7) | -1.6 (4.7) | -0.4 (9.2)
Statistical Analysis 1: Comparison: EBR/GZR vs SOF/LDV; RBV free EBR/GZR vs. SOF/LDV (all patients who started treatment by arm as treated); Test type: Superiority — Superiority test comparison based on whether the 95% CI includes zero; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.6 to 1.3] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

11. Primary Outcome: Median Change in Nausea PRO Score -Phase 1
Description: Patients completed the PROMIS® Nausea Short Form at Baseline (T1) and on-treatment. PROMIS raw scores from each of the completed questionnaires were converted to standardized T-scores. Change was calculated as the difference between baseline and on-treatment score. T-scores for the PROMIS Nausea and Vomiting 4a scale range from 45.0 - 80.1. Higher scores indicate worse nausea. Negative values for mean change represent improvement.
  The estimates of change and differences were obtained from a constrained longitudinal linear mixed-effects model that treated the baseline score as one of the outcomes.
Time Frame: Baseline to end of treatment
Population: Analysis limited to patients who completed baseline and on treatment Nausea short form during Phase 1 (up to last PrOD randomized) as treated.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg tablet): 1 - 3 tablets,1-2 times per day (dosage and duration per discretion of provider)
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
  RBV(Ribavirin) (200mg tablet): 1 - 3 tablets,1-2 times per day (dosage and duration per discretion of provider)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration as per discretion of HCV provider)
- PrOD With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  RBV(Ribavirin) (200mg tablet): 1 - 3 tablets,1-2 times per day (dosage and duration per discretion of provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 8 | 79 | 5 | 58 | 59 | 25
units on a scale | 0.4 [-6.5 to 10.0] | 0.0 [-22.2 to 20.8] | -6.1 [-8.0 to 0.9] | 0.0 [-21.6 to 23.7] | 0.0 [-19.2 to 22.2] | 0.0 [-25.2 to 31.7]

12. Primary Outcome: Median Change in Nausea PROMIS Score-EBR/GZR SOF/LDV
Description: Patients completed the PROMIS® Nausea Short Form at Baseline (T1) and on-treatment. PROMIS raw scores from each of the completed questionnaires were converted to standardized T-scores. Change was calculated as the difference between baseline and on-treatment score. T-scores for the PROMIS Nausea and Vomiting 4a scale range from 45.0 - 80.1. Higher scores indicate worse nausea. Negative values for change represent improvement.
  The estimates of change and differences were obtained from a constrained longitudinal linear mixed-effects model that treated the baseline score as one of the outcomes.
Time Frame: Baseline- On Treatment (up to 16 weeks)
Measure: Median (Full Range); unit: score on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) RBV(Ribavirin) (200mg tablet): 1 - 3 tablets,1-2 times per day (dosage and duration per discretion of provider)
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider) Ribavirin (RBV) 200 mg tablet: RBV(Ribavirin) (200mg tablet): 1 - 3 tablets,1-2 times per day (dosage and duration per discretion of provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 37 | 381 | 9 | 202
score on a scale | 0.0 [-21.0 to 18.3] | 0.0 [-29.2 to 23.3] | 0.0 [-8.0 to 7.3] | 0.0 [-26.1 to 24.9]

13. Primary Outcome: Mean Change in Fatigue PRO Score -Phase 1
Description: Fatigue severity collected from validated, Patient Reported Outcomes survey (PROs), 'PROMIS Fatigue Short Form'. PROMIS® T-scores were computated to compare difference between baseline value of PROMIS score to the highest (worst) score during treatment. Results presented as computated t-score from baseline to average of on Treatment Scores. A positive (+) score suggests improvements in functional well-being. A negative (-) PRO change score is suggestive of symptom improvement or lack of drug side effect. PROMIS Fatigue Score scale per question: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always with 7 questions for a total maximum score of 35.
Time Frame: Baseline to On-treatment
Population: Analysis limited to patients who completed baseline and at least one on-treatment Fatigue PRO survey during phase 1 as treated.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg tablet): 1 to 3 tablets, once or twice daily (dosage and duration per discretion of provider). Total daily dosage ranged from 200 to 1200 mg daily.
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
  RBV (Ribavirin) 200mg tablet: 1 to 3 tablets, once or twice daily at discretion of provider. Total daily dosage ranged from 200 to 1200 mg.
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
- PrOD With RBV: Patients received PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV).
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  RBV (200 mg tablet): 1-3 tablets, 1-2 times per day, daily for 12 to 24 weeks (dosage and duration at discretion of provider)
- PrOD: Patients received PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks without Ribavirin (RBV).
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 9 | 78 | 5 | 59 | 59 | 27
units on a scale | 1.5 (7.7) | -1.2 (9.2) | -7.2 (10.2) | -2.0 (7.9) | -1.9 (11.3) | -3.0 (7.9)
Statistical Analysis 1: Comparison: EBR/GZR vs PrOD; RBV free EBR/GZR vs. PrOD regimens as reported in PRO (all patients who started treatment by arm as treated, population is limited to as randomization date of the last PrOD patient start date). Analysis limited to RBV free regimen in consideration RBV usage determined by provider and not study randomization; Test type: Superiority — Superiority test based on whether the 95% CI includes zero; Mean Difference (Net) = 1.8, 95% CI 2-sided [-1.9 to 5.5] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method
Statistical Analysis 2: Comparison: SOF/LDV vs PrOD; RBV free SOF/LDV vs. PrOD regimens as reported in PRO (all patients who started treatment by arm as treated, population is limited to as randomization date of the last PrOD patient start date); Test type: Superiority — Superiority test based on whether the 95% CI includes zero; Mean Difference (Net) = -1.0, 95% CI 2-sided [-4.6 to 2.7] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

14. Primary Outcome: Mean Change in Fatigue PRO -EBR/GZR vs SOF/LDV
Description: as for outcome 13
Time Frame: Baseline and Average On-Treatment Score
Population: Patients with Baseline PROMIS Fatigue score who started treatment by arm as treated (Period 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV (at discretion of provider) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion)
  Ribavirin (RBV) 200 mg tablet: 1 - 3 tablets,1-2 times per day, daily for 12 to 16 weeks (dosage and duration per discretion of provider).
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) once daily without RBV (at discretion of provider) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion)
- SOF/LDV With RBV: Patients received sofosbuvir/ledipasvir orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food, daily for 12 - 24 weeks (use of RBV and dosage at discretion of provider)
- SOF/LDV: Patients received sofosbuvir/ledipasvir orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 38 | 398 | 10 | 213
score on a scale | -1.0 (7.7) | -2.1 (9.1) | -3.7 (8.3) | -2.2 (8.7)
Statistical Analysis 1: Comparison: EBR/GZR vs SOF/LDV; Analysis limited to RBV free regimens in consideration that RBV usage determined by provider and not study randomization. All patients who started treatment by arm as treated; Test type: Superiority — Superiority test comparison based on presence of zero in 95% CI; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.4 to 1.6] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

15. Primary Outcome: Median Change in Fatigue -Phase 1
Description: as for outcome 13
Time Frame: Baseline to End of Treatment
Population: Analysis is limited to patients who completed baseline and on-treatment fatigue PRO during Phase 1 (last PrOD patient started). Safety profiles of the evaluated regimens in PRIORITIZE are by actual treatment received.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EBR/GZR Regimen: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV With RBV: Patients received sofosbuvir/ledipasvir orally once daily with or without food 12 to 24 weeks with or without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- PrOD Regimen With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- PrOD: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks without Ribavirin (RBV).
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR Regimen | SOF/LDV With RBV | SOF/LDV | PrOD Regimen With RBV | PrOD
Number analyzed (Participants) | 9 | 78 | 5 | 59 | 59 | 27
units on a scale | 2.2 [-9.2 to 15.0] | -0.9 [-31.0 to 24.2] | -10.2 [-20.0 to 7.2] | -3.4 [-21.1 to 16.4] | -0.2 [-33.4 to 17.8] | -4.1 [-17.5 to 16.6]

16. Primary Outcome: Median Change in Fatigue-Phase 2
Description: as for outcome 13
Time Frame: Baseline-On Treatment (up to 16 weeks)
Population: Analysis limited to Period 2 -as treated, participants who completed baseline and on-treatment surveys.
Measure: Median (Full Range); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received elbasvir/grazoprevir (EBR/GZR) tablet orally once daily with or without Ribavirin (RBV) for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks Ribavirin (RBV) (200 mg tablet)- 1-3 tablets orally, once or twice daily (dosage at provider discretion). Total daily dosage 200 -1200 mg.
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (treatment duration per discretion of provider)
  sofosbuvir/ledipasvir: 1 Sofosbuvir/Ledipasvir (400/90 mg) tablet once daily with or without food for approximately 12 to 24 weeks Ribavirin (200 mg tablet): 1-3 tablets, once or twice daily (treatment duration and dosage of ribavirin as per discretion of HCV provider).
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 38 | 398 | 10 | 213
units on a scale | -1.3 [-19.1 to 15.0] | -1.2 [-31.6 to 24.2] | -2.4 [-20.0 to 7.2] | -1.4 [-39.0 to 20.7]

17. Primary Outcome: Mean Change in HCV- PRO- Phase 1
Description: HCV-PRO, a survey for patients with HCV that measures physical, emotional, and social functioning, productivity, intimacy, and perception of quality of life, was used to assess 'overall functioning and well-being'. In general, lower score is worst outcome and higher scores indicate greater well-being and functioning. However, for ease of interpretation, HCV-PRO scale has been transformed by using '100 - HCV-PRO' ultimately revising the score to mean 0 (lowest score) is best to 100 (worst outcome). A positive change (End of treatment to baseline) suggests improvements in functional well-being.
  Total score = (SUM-N)/(4*N)*100, where N is the number of questions answered.
Time Frame: Baseline to End of Treatment
Population: Analysis limited to patients who completed baseline and at least one on treatment Fatigue Short form. Evaluation is based on actual HCV regimen received.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV (at discretion of provider) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet orally once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dose ranging from 200 mg to 1200 mg.
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) once daily without RBV (at discretion of provider) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet orally once daily with or without food for 12 to 16 weeks (duration per provider discretion)
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration and use of ribavirin is per discretion of HCV provider)
- PrOD With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  RBV (200 mg tablet): 1-3 tablets, once or twice daily for 12 to 24 weeks (dosage and duration at discretion of provider).
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 9 | 84 | 5 | 61 | 61 | 29
units on a scale | -0.9 (12.4) | 5.6 (14.0) | 2.5 (7.1) | 6.9 (16.9) | 3.2 (22.8) | 9.9 (12.6)
Statistical Analysis 1: Comparison: EBR/GZR vs PrOD; Analysis based on RBV free regimens -all patients who started treatment by arm as treated, population is limited to as randomization date of the last PrOD patient start date; Test type: Superiority — Superiority test determined by comparing presence of zero in CI; Mean Difference (Net) = -4.3, 95% CI 2-sided [-9.9 to 1.3] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method
Statistical Analysis 2: Comparison: SOF/LDV vs PrOD; RBV free regimens as reported in PRO (all patients who started treatment by arm as treated, population limited to as randomization date of the last PrOD patient start date); Test type: Superiority — Superiority comparison by viewing presence of zero in CI; Mean Difference (Net) = 3.0, 95% CI 2-sided [-3.4 to 9.4]

18. Primary Outcome: Median Change in HCV-PRO (Overall Well Being) -Phase 1
Description: as for outcome 17
Time Frame: Baseline to End of Treatment
Population: Analysis limited to patients who completed baseline and at least one survey while on treatment up to end of treatment. Evaluation was based on actual regimen received versus regimen to which patient was randomized.
Measure: Median (Full Range); unit: score on a scale
Groups:
- EBR/GZR With RBV: Subjects will take EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg tablet): 1 to 3 tablets, once or twice daily (dosage and duration per discretion of provider)
- EBR/GZR: Subjects will take EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV 400/90 mg tablet: 1 tablet once daily for approximately 12 to 24 weeks (treatment duration as HCV provider discretion)
- PrOD With RBV: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV). Treatment duration and use of ribavirin as per HCV provider
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks (dosage at discretion of provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage ranging from 200 - 1200 mg.
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
Number analyzed (Participants) | 9 | 84 | 5 | 61 | 61 | 29
score on a scale | 0.0 [-21.9 to 16.4] | 4.3 [-32.8 to 43.0] | 4.7 [-9.4 to 7.8] | 4.7 [-39.8 to 47.7] | 3.1 [-50.0 to 71.9] | 8.6 [-19.7 to 31.3]

19. Primary Outcome: Mean Change in HCV-PRO (Functional Well-being) EBR/GZR vs. SOF/LDV Score-Phase 2
Description: HCV-PRO, a survey designed to assess functional status of patients with HCV and measures physical, emotional, and social functioning, productivity, intimacy, and perception of quality of life, was used to assess functional well-being. In general, lower score is worst outcome and higher scores indicate greater well-being and functioning. However, for ease of interpretation, HCV-PRO scale has been transformed by using '100 - HCV-PRO' ultimately revising the score to mean 0 (lowest score) is best to 100 (worst outcome). A positive change (End of treatment to baseline) suggests improvements in functional well-being.
  Total score = (SUM-N)/(4*N)*100, where N is the number of questions answered. End of Treatment -Baseline were used to calculate CHANGE in outcome. Number of subjects reflects participants from both Phase 1 and 2.
Time Frame: End of Treatment - Baseline
Population: Patients with completed Baseline and End of Treatment HCV-PRO survey who started treatment by arm as treated (Period 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV (at discretion of provider) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet orally once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dose ranging from 200 mg to 1200 mg.
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage ranged from 200 to 1200 mg.
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
Arm/Group | EBR/GZR With RBV | EBR/GZR | SOF/LDV With RBV | SOF/LDV
Number analyzed (Participants) | 40 | 413 | 10 | 226
score on a scale | 3.2 (18.6) | 6.1 (15.7) | 6.3 (10.7) | 6.8 (18.3)
Statistical Analysis 1: Comparison: EBR/GZR vs SOF/LDV; Analysis based on RBV free regimens in consideration that RBV usage was determined by provider and not study randomization. Population includes patients who started treatment by arm as treated; Test type: Superiority; Mean Difference (Net) = -0.7, 95% CI 2-sided [-3.6 to 2.1] — CI for mean derived from PROC TTEST, difference in mean and its 95%CI was calculated by Satterthwaite method

20. Primary Outcome: 16 Wk EBR/GZR With RBV Efficacy on Patients With HCV RASs
Description: Efficacy of Hepatitis C Virus (HCV) Treatment with Zepatier (Elbasvir/Grazobevir) with Ribavirin (RBV) for 16 weeks when used in Genotype 1a patients with Baseline RASs (NS5a Resistance Associated Substitutions or RAPs -Resistance Associated Polymorphisms).
  Efficacy defined as HCV RNA undetectable 12 weeks post treatment. Table excludes Genotype 1b patients.
Time Frame: 12 weeks post treatment
Population: All Genotype 1a patients who started treatment by arm randomized (Elbasvir/Grazobevir) with Baseline RAS at any location (28, 30, 31, or 93)
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR With RBV-16 Weeks: Subjects received EBR/GZR (elbasvir/grazoprevir) once daily with Ribavirin (RBV) for 16 weeks (as per provider discretion)
  EBR/GZR: Elbasvir/grazoprevir (50/100mg tablet) 1 tablet once daily with or without food
  RBV (200 mg tablet): 1-3 tablets once or twice daily for 16 weeks (dosage and duration at discretion of provider). Total dosage ranging from 200 mg to 1200 mg daily.
Arm/Group | EBR/GZR With RBV-16 Weeks
Number analyzed (Participants) | 38
Participants | 34

21. Secondary Outcome: Treatment Non-Adherence Probability Estimates
Description: The Voils Medication Adherence Survey (VMAS) was used to evaluate medication adherence during HCV treatment. Participants responded to three questions about the extent of adherence during the past seven days of treatment (during early and late on-treatment occasions). Participants responded using a five-point ordinal scale of missed dosing from 1 (none of the time) to 5 (all of the time). On each occasion participants were coded as being "Non-adherent" if any response was > 1, otherwise they were coded as "Adherent". Probability estimates of percentage of patients reporting non-adherence were calculated per HCV treatment (Direct Acting Antiviral-DAA) regimen: 1)EBR/GZV (elbasvir/grazoprevir, 2)SOF/LDV (sofosbuvir/ledipasvir), 3)PrOD
Time Frame: 12-16 weeks of HCV treatment
Population: Analysis is limited to participants to patients who started treatment prior to January 2017 (last day patient started on PrOD treatment)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with or without RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage ranging from 200-1200 mg.
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks with or without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- PrOD: PrOD -(ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with or without Ribavirin
  ombitasvir/paritaprevir/ritonavir (12.5/75/50mg tablet): 2 tablets once daily for 12 to 24 weeks (treatment duration as per HCV provider)
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks RBV (200 mg tablet): 1-3 tablets once or twice daily for 12 to 24 weeks (dosage and duration at discretion of provider)
Arm/Group | EBR/GZR | SOF/LDV | PrOD
Number analyzed (Participants) | 151 | 108 | 146
percentage of patients | 23 [17 to 29] | 19 [10 to 27] | 26 [19 to 33]

22. Secondary Outcome: Change in HCV-associated Symptoms (PROMIS Measures) After HCV Treatment Initiation
Description: Change in HCV-associated symptoms was calculated as the mean differences of mean scores from multiple surveys from the NIH Patient-Reported Outcomes Measurement Information System (PROMIS)-- Fatigue, nausea, belly pain, sleep disturbance, and diarrhea) and functional status (well-being) when comparing baseline to early post-treatment and late post treatment surveys. Mean change scores were calculated by comparing baseline to early post-treatment (1 yr) and late post-treatment (approximately 3 years) surveys. T-scores for the PROMIS Nausea and Vomiting 4a scale range from 45.0 - 80.1. Higher scores indicate worse nausea. Negative values for mean change represent improvement.Negative numbers suggest better symptoms (improvement in HCV-associated symptoms). PROMIS Fatigue Score scale per question: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always with 7 questions for a total maximum score of 35.HCV-PRO positive estimates suggest baseline functional well-being improvement.
Time Frame: 1 year post treatment discontinuation (Early post-tx)
Population: Analysis includes all patients who started treatment on either EBR/GZR or SOF/LDV regimen and is limited to patients who completed surveys. Analysis does not decipher between RBV usage given RBV usage was based on HCV provider selection and not study randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- EBR/GZR Regimen: Patients received elbasvir/grazoprevir tablet tablet once daily with or without RBV (at discretion of provider) for 12 to 16 weeks (provider discretion)
  elbasvir/grazoprevir: Elbasvir/grazoprevir (50/100mg) tablet once daily with food and with RBV: Ribavirin (200 mg/pill) 1-3 pills/day, 1-2 times/day. Total daily dosage ranged from 200 to 1200 mg.
- SOF/LDV Regimen: Patients received 1 tablet SOF/LDV(sofosbuvir/ledipasvir) orally once daily with or without ribavirin (RBV) (per discretion of provider) with or without food 12 to 24 weeks
  SOF/LDV/sofosbuvir/ledipasvir: Sofosbuvir/Ledipasvir (400/90 mg) for approximately 12 to 24 weeks (treatment duration is per discretion of HCV provider) RBV: Ribavirin (200mg pill) 1-3 pills, once or twice/day -dosage at discretion of provider. Total daily dosage ranged from 200 to 1200 mg.
Arm/Group | EBR/GZR Regimen | SOF/LDV Regimen
Number analyzed (Participants) | 507 | 286
units on a scale
  Nausea: number analyzed (Participants) | 505 | 285
  Nausea | 0.00 [-2.34 to 2.35] | -4.99 [-8.16 to -1.81]
  Belly Pain: number analyzed (Participants) | 503 | 283
  Belly Pain | -0.82 [-3.52 to 1.87] | -6.47 [-10.09 to -2.84]
  Diarrhea: number analyzed (Participants) | 504 | 282
  Diarrhea | -1.12 [-3.46 to 1.22] | -5.77 [-8.91 to -2.64]
  Fatigue: number analyzed (Participants) | 506 | 285
  Fatigue | -2.08 [-4.74 to 0.58] | -7.59 [-11.17 to -4.01]
  Sleep Disturbance: number analyzed (Participants) | 505 | 283
  Sleep Disturbance | 0.65 [-0.70 to 2.00] | -1.72 [-3.81 to 0.37]
  Cognitive Impairment: number analyzed (Participants) | 507 | 282
  Cognitive Impairment | -0.54 [-2.43 to 1.35] | -4.48 [-7.12 to -1.83]
  HCV-PRO | 8.02 [3.94 to 12.11] | 9.90 [4.27 to 15.52]

23. Secondary Outcome: Post-treatment Progression/Regression of Liver Disease-Fib-4
Description: Mean change (delta) in FIB-4, an indirect non-invasive measure of liver fibrosis, calculated as baseline median -long term follow up median, following SVR after any of the study treatment regimens. Change in FIB-4 where negative values indicate improvement in liver fibrosis score and positive values indicate worsening of fibrosis score. There is no upper or lower limit for change. FIB-4 = age (years) * AST(IU/L)/Platelets (10^3/L) * ALT^.5(IU/L). In general, Score of 0-1.29 is low risk for advanced fibrosis, 1.30-1.67: intermediate risk for advanced liver fibrosis, >2.67: high risk for advanced fibrosis.
Time Frame: Baseline to up to 3 years post treatment discontinuation
Population: Population analyzed limited to cirrhotic patients who had two separate FIB-4 values collected as part of standard care and achieved SVR (defined as undetectable HCV 24 weeks post treatment). Given pragmatic trial design, availability of fibrosis markers is limited thereby restricting analysis (substantially limited sample size) to difference in fibrosis markers following SVR with any HCV treatment used in study.
Measure: Median (Full Range); unit: score on a scale
Groups:
- EBR/GZR, SOF/LDV or PrOD Based HCV Treatment: Elbasvir/grazoprevir (EBR/GZR): (50/100mg) tablet once daily with food for 12 to 16 weeks with or without RBV (Ribavirin usage as per provider discretion).
  Sofosbuvir/ledipasvir (SOF/LDV)/ (400/90 mg) 1 tablet once daily for approximately 12 to 24 weeks (treatment duration is per discretion of HCV provider) with or without RBV (RBV usage as per provider discretion):
  PrOD: Two ombitasvir/paritaprevir/ritonavir once daily and dasabuvir twice daily for 12 to 24 weeks + RBV (provider discretion)
  ombitasvir/paritaprevir/ritonavir (Phase 1 only): (Phase 1 only) Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg) for 12 to 24 weeks (treatment duration and use of ribavirin as per HCV provider)
  Dasabuvir: 250 mg daily for 12 to 24 weeks RBV: Ribavirin 200 to 600 mg once or twice daily RBV (Ribavirin)- 200mg pill, 1-3 pills/day once or twice daily (use and dosing per discretion of HCV provider).
Arm/Group | EBR/GZR, SOF/LDV or PrOD Based HCV Treatment
Number analyzed (Participants) | 108
score on a scale | -1.36 [-11.02 to 10.67]

24. Secondary Outcome: Change in Functional Status (HCV-PRO) Within Treatment
Description: HCV-PRO score, a validated PROMIS survey used to evaluate overall functioning and well-being in HCV patients, was utilized to compare long-term 'within treatment' changes of functional well-being. In general, lower score is worst outcome and higher scores indicate greater well-being and functioning. However, for ease of interpretation, HCV-PRO scale has been transformed by using '100 - HCV-PRO' ultimately revising the score to mean 0 (lowest score) is best to 100 (worst outcome). A positive estimate (Post treatment to baseline) suggests baseline functional well-being improvement.
  Total score = (SUM-N)/(4*N)*100, where N is the number of questions answered.
Time Frame: Treatment start date up to 2 years post-treatment
Population: Analysis limited to patients who completed HCV-PRO assessments during post-treatment. For this safety analysis, regimen is based on treatment received versus treatment to which patient was randomized. Arms with and without RBV are combined in consideration that usage of RBV was decided by HCV provider and not part of study randomization.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- EBR/GZR Regimen: Subjects will take EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with or without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg to 600mg tablet): 1 to 3 tablets once or twice daily (dosage and duration per discretion of provider)
- SOF/LDV Regimen: Subjects will take 1 tablet SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with or without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
Arm/Group | EBR/GZR Regimen | SOF/LDV Regimen
Number analyzed (Participants) | 498 | 295
score on a scale
  9 months post treatment | 8.02 [3.94 to 12.11] | 9.90 [4.27 to 15.52]
  20 months post treatment | 9.87 [5.48 to 14.27] | 11.54 [5.07 to 18.02]

25. Secondary Outcome: Number of Participants With Adverse Events That Caused Treatment Discontinuation-EBR/GZR vs. LDV/SOF
Description: The number of participants with adverse events that led to early treatment discontinuation (defined as duration less than originally prescribed treatment regimen)
Time Frame: Treatment start date through treatment completion (up to 24 weeks)
Population: As randomized and treated population during Phase 1 and 2 (See Period 1). Analysis based on HCV DAA regimen randomization per study. Differentiation between RBV usage was not included in analysis given that RBV was not part of study randomization but rather decided by HCV provider.
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR Regimen: Patients received EBR/GZR (elbasvir/grazoprevir ) tablet once daily for 12 to 16 weeks (duration of treatment per provider discretion) with or without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg to 600mg pill): 1 to 3 pill once or twice daily (dosage and duration per discretion of provider)
- SOF/LDV Regimen: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with or without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg pill: 1 to 3 pills once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage ranged from 200 to 1200 mg.
Arm/Group | EBR/GZR Regimen | SOF/LDV Regimen
Number analyzed (Participants) | 700 | 428
Participants | 12 | 4

26. Secondary Outcome: HCV SVR Durability -No Cirrhosis
Description: Number/Percentage of patients with persistence of viral cure, SVR (SVR = Sustained Virologic Response)- defined as undetectable HCV RNA at least 24 weeks following HCV Treatment.
Time Frame: 24 weeks post-end of treatment up to 153 weeks
Population: Analysis limited to patients who have HCV RNA result at least 24 weeks after end of treatment regimen as per period 1 (As randomized).
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR: Patients received EBR/GZV tablet (elbasvir/grazoprevir) once daily for 12 to 16 weeks
  EBR/GZV (50/100mg) tablet: 1 tablet once daily with or without food 12 to 16 weeks
- EBR/GZR With Ribavirin: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets, once or twice daily orally with food (use of RBV and dosage at discretion of provider). Total daily dosage ranged from 200 to 1200 mg.
Arm/Group | EBR/GZR | EBR/GZR With Ribavirin | SOF/LDV | SOF/LDV With RBV | PrOD | PrOD With RBV
Number analyzed (Participants) | 255 | 17 | 146 | 2 | 14 | 36
Participants | 255 | 17 | 146 | 2 | 14 | 36

27. Secondary Outcome: HCV SVR Durability-Patients With Cirrhosis
Description: Percentage of Cirrhotic patients with persistence of viral cure, SVR, (SVR= Sustained Virologic Response) defined as undetectable HCV RNA at least 24 weeks following HCV Treatment.
Time Frame: Up to 132 weeks post HCV treatment
Population: Analysis limited to patients who had HCV viral load result at least 24 weeks after treatment and analyzed as per randomized (Period 1)
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir) once daily with RBV (Ribavirin) for 12 to 16 weeks
  EBR/GZR (50/100mg tablet): 1 tablet once daily with or without food for 12 to 16 weeks (duration per provider discretion) Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
Arm/Group | EBR/GZR | EBR/GZR With RBV | SOF/LDV | SOF/LDV With RBV | PrOD | PrOD With RBV
Number analyzed (Participants) | 43 | 7 | 35 | 7 | 6 | 7
Participants | 43 | 7 | 35 | 7 | 6 | 7

28. Secondary Outcome: Impact of Baseline NS5A RASs on Treatment Outcomes-Phase 2
Description: Number of participants who achieved SVR (sustained virologic response), defined as undetectable HCV RNA 12 weeks post-treatment with RASs (Resistant Associated Substitutions) after treatment with EBR/GZR or SOF/LDV regimen
Time Frame: 12 weeks post HCV treatment
Population: Analysis is based on as assigned by randomization and patients with available RAS data. Exploratory RAS analysis is grouped by DAA regimen with or without RBV given 1)RBV usage was decided by HCV provider and not part of study randomization and small sample size (limited number of RAS in regimens with RBV)
Measure: Count of Participants; unit: Participants
Groups:
- EBR/GZR Regimen: Patients received EBR/GZR (elbasvir/grazoprevir) once daily for 12 to 16 weeks (duration of treatment per provider discretion) with or without Ribavirin (RBV) (per provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food for 12 to 16 weeks
  RBV(Ribavirin) (200mg to 600mg tablet): 1 to 3 tablets once or twice daily (usage, dosage and duration per discretion of provider) (Total dosage ranging from 200 mg to 1200 mg daily)
- SOF/LDV Regimen: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily 12 to 24 weeks (per discretion of provider) with or without ribavirin (RBV) (per discretion of provider)
  SOF/LDV (400/90 mg tablet): 1 tablet once daily with or without food for approximately 12 to 24 weeks (treatment duration per discretion of HCV provider)
  Ribavirin (RBV) 200 mg tablet: 1 to 3 tablets once or twice daily orally with food (use of RBV and dosage at discretion of provider)
Arm/Group | EBR/GZR Regimen | SOF/LDV Regimen
Number analyzed (Participants) | 560 | 337
Participants
  With NS5a RAS: number analyzed (Participants) | 54 | 47
  With NS5a RAS | 47 | 42
  Without NS5a RAS: number analyzed (Participants) | 506 | 290
  Without NS5a RAS | 485 | 286
Statistical Analysis 1: Comparison: EBR/GZR Regimen vs SOF/LDV Regimen; Test type: Equivalence — Pre-specified equivalence range +/-5%; Mean Difference (Net) = -2.3, 95% CI 2-sided [-15.3 to 11.3]

ADVERSE EVENTS:
Time Frame: 28 weeks. Adverse events collected up until final viral outcome is determined (approximately 12 weeks after HCV treatment completion).
Description: An adverse event (AE) is any untoward medical occurrence abstracted from the submitted patient medical records. In order to evaluate the safety profiles of the evaluated regimens, all safety analyses were performed based on 'actual treatment received' (as described in Period 2) rather than treatment to which subject was 'randomized'
Groups:
- EBR/GZR: Patients received EBR/GZR (elbasvir/grazoprevir) tablet once daily without RBV for 12 to 16 weeks (provider discretion)
  EBR/GZR: Elbasvir/grazoprevir (50/100mg tablet) 1 tablet once daily with or without food
- EBR/GZR With RBV: Patients received EBR/GZR (elbasvir/grazoprevir tablet) tablet once daily with Ribavirin (RBV) for 12 to 16 weeks (provider discretion)
  EBR/GZR (Elbasvir/grazoprevir) 50/100mg tablet: 1 tablet once daily with or without food with RBV (200 to 600 mg once or twice daily) for 12 to 16 weeks
- SOF/LDV With RBV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks with ribavirin (RBV) (per discretion of provider)
  SOF/LDV (Sofosbuvir/Ledipasvir) (400/90 mg tablet) 1 tablet taken daily for approximately 12 to 24 weeks with RBV (Ribavirin) 200 mg: 1-3 pills, one to two times daily (dosage at discretion of HCV provider). Total daily dosage ranged fro 200 to 1200 mg.
- SOF/LDV: Patients received SOF/LDV (sofosbuvir/ledipasvir) orally once daily with or without food 12 to 24 weeks (treatment duration per discretion of provider)
  SOF/LDV (Sofosbuvir/Ledipasvir )(400/90 mg tablet) 1 tablet orally taken daily for approximately 12 to 24 weeks
- PrOD With RBV: PrOD (ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks with Ribavirin (RBV) (treatment at duration provider discretion)
  ombitasvir/paritaprevir/ritonavir: 2 tablets orally once daily (12.5/75/50mg) for 12 to 24 weeks
  Dasabuvir (250 mg tablet): 1 tablet orally once or twice daily for 12 to 24 weeks Ribavirin (200 mg pill): 200 to 600 mg once or twice daily (dosage at provider discretion). Total daily dosage ranged from 200 to 1200 mg.
- PrOD: Patients received PrOD orally (ombitasvir/paritaprevir/ritonavir and dasabuvir) daily for 12 to 24 weeks without Ribavirin (RBV) (provider discretion)
  Ombitasvir/paritaprevir/ritonavir (12.5/75/50mg): 2 tablets taken once orally daily for 12 to 24 weeks (treatment duration as per HCV provider)
  Dasabuvir (250 mg tablet): 1 tablet once or twice daily for 12 to 24 weeks
Arm/Group | EBR/GZR | EBR/GZR With RBV | SOF/LDV With RBV | SOF/LDV | PrOD With RBV | PrOD
All-Cause Mortality (participants affected / at risk) | 6/664 | 0/56 | 0/15 | 4/394 | 1/99 | 0/47
Serious Adverse Events (participants affected / at risk) | 30/664 | 2/56 | 0/15 | 6/394 | 5/99 | 0/47
Other Adverse Events (participants affected / at risk) | 298/664 | 46/56 | 8/15 | 184/394 | 74/99 | 32/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBR/GZR (N=664) | EBR/GZR With RBV (N=56) | SOF/LDV With RBV (N=15) | SOF/LDV (N=394) | PrOD With RBV (N=99) | PrOD (N=47)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal Syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Detoxification (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Gastric ulcer perforation
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status change (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Hematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBR/GZR (N=664) | EBR/GZR With RBV (N=56) | SOF/LDV With RBV (N=15) | SOF/LDV (N=394) | PrOD With RBV (N=99) | PrOD (N=47)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 17 (17) | 2 (2) | 0 (0) | 20 (20) | 0 (0) — Anemia
Abdominal discomfort (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 15 (15) | 7 (7) | 0 (0) | 11 (11) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8) | 0 (0) | 11 (11) | 9 (9) | 1 (1) — Dyspnea
Fatigue (Nervous system disorders) | 105 (105) | 18 (18) | 5 (5) | 82 (82) | 35 (35) | 5 (5)
Headache (Nervous system disorders) | 94 (94) | 12 (12) | 1 (1) | 68 (68) | 15 (15) | 9 (9)
Insomnia (Nervous system disorders) | 26 (26) | 6 (6) | 1 (1) | 10 (10) | 8 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 54 (54) | 12 (12) | 3 (3) | 34 (34) | 23 (23) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 45 (45) | 3 (3) | 2 (2) | 19 (19) | 5 (5) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 11 (11) | 5 (5) | 1 (1) | 11 (11) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 3 (3) | 0 (0) | 12 (12) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (16) | 5 (5) | 0 (0) | 12 (12) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 3 (3) | 0 (0) | 14 (14) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (Infections and infestations) | 18 (18) | 3 (3) | 0 (0) | 7 (7) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 13 (13) | 3 (3) | 0 (0) | 13 (13) | 8 (8) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 8 (8) | 2 (2) | 1 (1) | 9 (9) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 1 (1) | 1 (1) | 13 (13) | 4 (4) | 0 (0)
Chest Pain (Cardiac disorders) | 10 (10) | 1 (1) | 1 (1) | 9 (9) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Gastrointestinal disorders) | 9 (9) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Oedema Peripheral (Vascular disorders) | 12 (12) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) — Peripheral edema Edema Peripheral
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This pragmatic trial allowed patients who were randomized to SOF/LDV but unable to obtain SOF/LDV (due to limitations in access from insurance, etc.) to be treated with the accessible, alternative DAA regimens. This contributed to the variance from 'as randomized' population to the 'as treated' population. Rapidly changing HCV landscape led to discontinuation of PrOD treatment regimen and modification of initial analysis plan including reduction of original sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02786537/Prot_SAP_000.pdf